CLINICAL TRIAL: NCT00694447
Title: Exploring Outcomes and Mechanisms of Acupuncture in Treating Pain and Sleep Disturbance in Knee Osteoarthritis
Brief Title: Acupuncture for Pain and Sleep Disturbance in Knee Osteoarthritis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: Southeast Center of Excellence in Geriatric Medicine (Unknown); The John A. Hartford Foundation (Other)
Responsible Party: Principal Investigator, Wei Huang MD, PhD, Principal Investigator, Emory University
Other Study IDs: IRB00000143; Grant #97333-G
Record Dates: First submitted 2008-06-06; First posted 2008-06-10 (Estimated); Last update posted 2013-11-21 (Estimated); Status verified 2013-11

CONDITIONS: Sleep; Pain
MeSH Terms: conditions — Pain | interventions — Acupuncture Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Real acupuncture (Experimental): Real acupuncture
  Interventions: Procedure: Acupuncture
- Sham acupuncture (Sham Comparator): Sham acupuncture
  Interventions: Procedure: Acupuncture

INTERVENTIONS:
Procedure: Acupuncture

SUMMARY:
The hypotheses of this study are: In the older population with knee OA,

* When acupoints are chosen for both sleep and pain, there are additive effects on sleep improvement and pain relief (i.e. no interaction).
* Main effects of acupuncture on sleep improvement and pain relief are anticipated when acupoints are separately targeted for sleep and for pain, respectively.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with knee osteoarthritis, diagnosed by the ACR clinical diagnosis criteria for idiopathic OA, with at least Kellgren and Lawrence grading II and above. AND,
2. Present with knee pain at least half of the time. AND,
3. Complain of sleep disturbances associated with knee OA, with Pittsburgh Sleep Quality Index > 5 [36].

Exclusion Criteria:

1. Patients with diagnosis of obstructive sleep apnea (OSA). OR,
2. Patients with dense hemiplegia secondary to cerebrovascular accident. OR,
3. NYHA Class III - patients with heart failure condition limited by minimal activity. OR,
4. Severe COPD with shortness of breath at minimal exertion. OR,
5. Peripheral vascular disease with severe claudication. OR,
6. Dementia with Mini Mental Status Exam score of 20 or less. OR,
7. Patients who received knee intra-articular corticosteroid injection within 4 weeks prior to the study or who received acupuncture treatment within 6 months. OR,
8. Unwilling to come off narcotic pain medication. OR,
9. History of bleeding diathesis or currently on anticoagulation. OR,
10. Patients currently engaged in medical legal cases related to OA or disability.

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2007-02; Primary Completion 2008-04 (Actual)

PRIMARY OUTCOMES:
Sleep disturbances as recorded by wrist actigraph, including sleep duration and sleep efficiency. Pain as measured by 0-10 VAS and WOMAC pain scores. | at least 3 months

SECONDARY OUTCOMES:
WOMAC disability scores, IDEEA gait patterns and activity levels, medication type and amount consumed, side effects, and medical care utilization. | at least 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Wei Huang, MD, PhD, Principal Investigator — Emory University
Locations (1):
- Wesley Woods Geriatric Hospital, Atlanta, Georgia, United States

REFERENCES:
- See also: publication from this study — http://onlinelibrary.wiley.com/doi/10.1111/j.1532-5415.2010.02886.x/abstract